CLINICAL TRIAL: NCT01390675
Title: Anesthesia for Catheter Aortic Valve ImplantATIOn Registry
Acronym: AVIATOR
Status: Recruiting | Type: Observational
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Principal Investigator, N Patrick Mayr, MD, Deutsches Herzzentrum Muenchen
Other Study IDs: GE DHM-AN-OR-2011/04; GE DHM-AN-OR-2011/04 (Other: Deutsches Herzzentrum München)
Record Dates: First submitted 2011-06-27; First posted 2011-07-11 (Estimated); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure; Excessive Amount of Blood / Fluid Transfusion; Intraoperative Cardiac Arrest During Cardiac Surgery; Critical Incident; Anesthesia; Failed Conscious Sedation During Procedure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In modern cardiac surgery and cardiology Transcatheter Aortic Valve Implantation (TAVI) is an emerging procedure for high-risk patients that are assumed to be otherwise inoperable. The investigators want to evaluate the specific intraoperative anesthesiologic characteristics cardiac anesthesiologists have to face during these procedures.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing transcatheter aortic valve implantation (TAVI)

Exclusion Criteria:

- Refusal by patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing transcatheter aortic valve implantation (TAVI)
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2011-06; Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Perioperative Care | 1 day
  major critical adverse events

SECONDARY OUTCOMES:
Up to 10 years | 10 Years
  all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Patrick N Mayr, M.D., Principal Investigator — Deutsches Herzzentrum München, Technische Universität München; Michael Joner, MD, Prof., Principal Investigator — Deutsches Herzzentrum München, Technische Universität München
Locations (1):
- Deutsches Herzzentrum München, Department of Anaesthesiology, Technische Universität München, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Mayr NP, Wiesner G, van der Starre P, Hapfelmeier A, Goppel G, Kasel AM, Hengstenberg C, Husser O, Schunkert H, Tassani-Prell P. Dexmedetomidine versus propofol-opioid for sedation in transcatheter aortic valve implantation patients: a retrospective analysis of periprocedural gas exchange and hemodynamic support. Can J Anaesth. 2018 Jun;65(6):647-657. doi: 10.1007/s12630-018-1092-4. Epub 2018 Feb 20. PMID 29464420